CLINICAL TRIAL: NCT01503242
Title: A Phase I Study of 90Y-BC8-DOTA Monoclonal Antibody, Fludarabine and TBI Followed by HLA-Matched, Allogeneic Peripheral Blood Stem Cell Transplant for the Treatment of Multiple Myeloma
Brief Title: 90 Y-BC8-DOTA Monoclonal Antibody, Fludarabine Phosphate, and Total-Body Irradiation Followed by Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2450.00; NCI-2010-02041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2450; 2450.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); R21CA155911 (NIH)
Record Dates: First submitted 2011-12-30; First posted 2012-01-02 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (monoclonal antibody, chemo, TBI, transplant) (Experimental): Patients receive 90Y-BC8 Ab IV on day -12 and fludarabine phosphate IV on days -4 to -2. Patients undergo TBI and allogeneic peripheral blood stem cell transplant on day 0. Patients also receive graft-vs-host disease prophylaxis comprising cyclosporine PO BID on days -3 to 56 with taper to day 180 or on days -3 to 100 with taper to 180; and mycophenolate mofetil IV or PO BID on days 0-27, or 0-40 with taper to 96.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Radiation: Total-Body Irradiation; Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation
Radiation: Yttrium Y 90 Anti-CD45 Monoclonal Antibody BC8 — Given IV
  Other Names: 90Y Anti-CD45 MoAb BC8

SUMMARY:
This phase I trial studies the side effects and best dose of yttrium Y 90 anti-CD45 monoclonal antibody BC8 when given together with fludarabine phosphate and total-body irradiation followed by donor peripheral blood stem cell transplant in treating patients with multiple myeloma. Radiolabeled monoclonal antibodies, such as yttrium Y 90 anti-CD45 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. Giving chemotherapy drugs, such as fludarabine phosphate, and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving yttrium Y 90 anti-CD45 monoclonal antibody BC8, fludarabine phosphate, and total-body irradiation before the transplant together with cyclosporine and mycophenolate mofetil after the transplant may stop this from happening and may be an effective treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the tissue localization of 111In-BC8-DOTA antibody therapy (Ab) and establish reproducibly favorable biodistribution.

II. To estimate the maximum tolerated dose (MTD) of radiation delivered via 90Y-BC8-DOTA Ab when combined with fludarabine phosphate (FLU) and 2 Gy total-body irradiation (TBI) as a preparative regimen followed by human leukocyte antigen (HLA)-matched, related or unrelated hematopoietic cell transplant (HCT) for patients with multiple myeloma.

SECONDARY OBJECTIVES:

I. To assess the potential efficacy of this approach, within the limits of a phase I study, by examining disease response, duration of remission, disease free survival (DFS), and overall survival (OS).

OUTLINE: This is a dose-escalation study of yttrium Y 90 anti-CD45 monoclonal antibody BC8 (90Y-BC8 Ab).

Patients receive 90Y-BC8 Ab intravenously (IV) on day -12 and fludarabine phosphate IV on days -4 to -2. Patients undergo TBI and allogeneic peripheral blood stem cell transplant on day 0. Patients also receive graft-vs-host disease prophylaxis comprising cyclosporine orally (PO) twice daily (BID) on days -3 to 56 with taper to day 180 or on days -3 to 100 with taper to 180; and mycophenolate mofetil IV or PO BID on days 0-27, or 0-40 with taper to 96.

After completion of study treatment, patients are followed up every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have history of symptomatic myeloma requiring treatment and meet one of the following requirements:

  * Have at least 1 high risk feature at diagnosis (including deletion 13 or hypodiploidy by conventional cytogenetics, t(4;14), t(14;16) or deletion 17 by fluorescence in situ hybridization [FISH], beta 2 microglobulin > 3.5, lactate dehydrogenase [LDH] greater than 1.5 x upper limit of normal [ULN], history of plasma cell leukemia) (prior to chemotherapy); OR
  * Have progressive disease on primary therapy with or without prior autologous stem cell transplant; OR
  * Have persistent or progressive disease following autologous transplant; it is acceptable for these patients to have a second transplant for disease reduction
* Bone marrow cellularity of >= 50% of age defined normal values by core biopsy; cellularity must be evaluated within 90 days of the dosimetry infusion and at least 21 days after receiving any cytoreductive/myelosuppressive chemotherapy
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Measured creatinine clearance > 50 ml/min or estimated creatinine clearance > 50 ml/min
* For females of childbearing potential, must have a negative pregnancy test
* Patients must have a human leukocyte antigen (HLA)-matched related donor or an unrelated donor who meets standard Seattle Cancer Care Alliance (SCCA) and or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) donation, or bone marrow donation as follows:

  * Related donor related to the patient and genotypically or phenotypically identical for HLA-A, B, C, DRB1 and DQB1; phenotypic identity must be confirmed by high-resolution typing
  * Unrelated donor:

    * Matched for HLA-A, B, C, DRB1 DQB1 by high resolution typing; OR
    * Mismatched for a single allele without antigen mismatching at HLA-A, B, or C as defined by high resolution typing but otherwise matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing
    * Patient and donor pairs homozygous at a mismatched allele, in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
  * Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA Class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* Ability to provide informed consent
* DONOR: Patients must have an HLA matched donor as well as standard Seattle Cancer Care Alliance (SCCA) and or National Marrow Donor Program (NMDP)/other donor center criteria for PBSC donation
* DONOR: Donors must consent and be eligible to undergo granulocyte colony-stimulating factor (GCSF) mobilization and PBSC harvest; marrow is not allowed as a source of stem cells on this study

Exclusion Criteria:

* Patients with the following organ dysfunction:

  * Left ventricular ejection fraction < 35%
  * Corrected diffusion capacity of carbon monoxide (DLCO) < 35% or receiving supplemental continuous oxygen
  * Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidences by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis, or symptomatic biliary disease
* Pregnant or breast-feeding females
* Circulating antibody against mouse immunoglobulin (HAMA)
* Prior allogeneic transplant
* Plasmacytomas > 1 cm in marrow areas measured by magnetic resonance imaging (MRI) or extramedullary plasmacytomas (radiated lesions are exempt from this criteria); patients may receive cytoreductive therapy, including allogeneic stem cell transplant (ASCT) (if high risk) or second ASCT (if failed a prior ASCT) to achieve disease control, but may not receive any cytoreductive therapy within 30 days of the dosimetry infusion and must have bone marrow cellularity meeting inclusion criteria obtained at least 21 days after any cytoreductive/myelosuppressive chemotherapy was last administered
* Prior radiation to maximally tolerated levels to any critical normal organ, or > 20 Gy prior radiation to large areas of the bone marrow (e.g., external radiation therapy to whole pelvis)
* Patients who are known to be seropositive for human immunodeficiency virus (HIV)
* Fertile men and women unwilling to use contraceptives during and for 12 months post-transplant
* Active central nervous system (CNS) disease at the time of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
MTD of radiation delivered via 90 Y-BC8-DOTA | Up to 180 days
  MTD is defined as the dose that is associated with a true dose-limiting toxicity (DLT) rate of 25%, where a DLT is defined as a grade III/IV regimen-related toxicity (Bearman scale) occurring within 30 days post-transplant. A two-parameter logistic model will be fit to the data, thereby generating a dose-response curve based on the observed toxicity rate at the various dose levels. Based on this fitted model, the MTD is estimated to be the dose that is associated with a toxicity rate of 25%.
Tissue localization of 111In-BC8-DOTA Ab | Up to 72 hours post infusion

SECONDARY OUTCOMES:
Disease response | Up to 3 years
Disease-free survival | Up to 3 years
Duration of remission | Up to 3 years
Overall survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Damian Green, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Tuazon SA, Sandmaier BM, Gooley TA, Fisher DR, Holmberg LA, Becker PS, Lundberg SJ, Orozco JJ, Gopal AK, Till BG, Coffey DG, Nartea ME, Matesan MC, Pagel JM, Rajendran JG, Press OW, Bensinger WI, Green DJ. 90Y-labeled anti-CD45 antibody allogeneic hematopoietic cell transplantation for high-risk multiple myeloma. Bone Marrow Transplant. 2021 Jan;56(1):202-209. doi: 10.1038/s41409-020-01000-3. Epub 2020 Jul 24. PMID 32710011